CLINICAL TRIAL: NCT03391648
Title: Incidence of Anesthesia-related Adverse Events and Obstetric Complications After Cesarean Delivery: a Retrospective Study
Brief Title: Incidence of Anesthesia-related Adverse Events and Obstetric Complications After Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kuo-Chen Chang, Attending physician, Far Eastern Memorial Hospital
Other Study IDs: 106116-E
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Adverse Effect, in Labor and Delivery
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cesarean
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation only

SUMMARY:
Recruit the parturients who underwent cesarean delivery at Far Eastern MemorialHospital during 2012-2016. After reviewing medical record related to the pregnancy, demographic data, prenatal exam, laboratory data, indication for cesarean section, perioperative events, etc. will be recorded. Analysis will be focused on incidence, temporal trend, and risk factors of anesthesia-related adverse events and obstetric complications.

ELIGIBILITY:
Inclusion Criteria:

* all parturients underwent cesarean section at Far Eastern Memorial Hospital during 2012-2016

Exclusion Criteria:

* missing data can't be collect during medical chart review

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parturients who undergo cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of anesthesia-related adverse events | Within 42 days after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No